CLINICAL TRIAL: NCT02680756
Title: A Phase 3b, Randomized, Controlled, Multicentre Study With Oral Ferric Maltol (Feraccru) or Intravenous Iron (Ferric Carboxy Maltose; FCM), for the Treatment of Iron Deficiency Anaemia in Subjects With Inflammatory Bowel Disease
Brief Title: Safety and Efficacy Study of Oral Ferric Maltol Compared to Intravenous Iron To Treat Iron Deficiency Anaemia in IBD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shield Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST10-01-304
Record Dates: First submitted 2016-02-09; First posted 2016-02-11 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Anemia, Iron-Deficiency; Inflammatory Bowel Disease; Crohn's Disease
Keywords: Iron Deficiency; Anaemia; Crohn's Disease; Deficiency Diseases; Inflammatory Bowel Diseases; Intestinal Diseases
MeSH Terms: conditions — Anemia, Iron-Deficiency; Inflammatory Bowel Diseases; Crohn Disease; Iron Deficiencies; Anemia; Deficiency Diseases; Intestinal Diseases | interventions — ferric maltol; ferric trimaltol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral ferric iron compound (Experimental): 30 mg capsules to be taken orally twice a day for 52 weeks
  Interventions: Drug: Ferric Maltol
- Intravenous iron (Active Comparator): Administered as per the local summary of product characteristics (SPC)
  Interventions: Drug: Ferric Carboxy Maltose

INTERVENTIONS:
Drug: Ferric Maltol
  Other Names: Feraccru; Ferric Trimaltol; ST10; ST10-01
  Arms: Oral ferric iron compound
Drug: Ferric Carboxy Maltose
  Arms: Intravenous iron

SUMMARY:
The purpose of this study is to compare the efficacy of ferric maltol and intravenous iron (IVI) Ferric Carboxy Maltose in the treatment of iron deficiency anaemia (IDA) and subsequent maintenance of haemoglobin in subjects with Inflammatory Bowel Disease (IBD).

DETAILED DESCRIPTION:
A phase 3b, randomized, controlled, multicentre study with oral ferric maltol or intravenous iron (FCM), for the treatment of iron deficiency anaemia in subjects with inflammatory bowel disease.

Approximately 242 eligible subjects will be randomised (1:1) to receive one of the following treatments for the duration of the study treatment period (52 weeks):

* Oral ferric maltol, 30 mg capsule bid.
* Intravenous iron (ferric carboxy maltose) as per SPC

In the FCM arm IV iron treatment will be repeated if the subject is iron deficient at any of the study visits.

Subject participation in the study will consist of 3 periods:

* Screening: Up to 14 days
* Randomised Treatment: 52 weeks
* Post-treatment safety follow-up: 14 days after study medication discontinuation

Primary efficacy and safety of ferric maltol and Intravenous iron (ferric carboxy maltose) will be evaluated after the first 12 weeks.

End of study evaluations will occur at Week 52 or premature discontinuation.

ELIGIBILITY:
All of the following criteria must be met to randomize a subject in the study:

1. Subjects must be competent to understand the information given in the Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved informed consent form and must sign and date the informed consent prior to any study mandated procedure
2. Subjects must be willing and able to comply with study requirements
3. Age ≥ 18 years
4. Subjects must have a confirmed diagnosis of IBD (endoscopic and/or biopsy)
5. Subjects must be considered suitable for intravenous iron treatment by the Investigator
6. Subjects must have iron deficiency anaemia defined by the following criteria:

   1. Hb 8.0 g/dL and ≤11.0 g/dL for women OR a Hb 8.0 g/dL and ≤12.0 g/dL for men
   2. AND Ferritin <30ng/ml OR Ferritin <100 ng/ml WITH Transferrin saturation (TSAT) <20%
7. Female subjects of childbearing potential (including perimenopausal females who have had a menstrual period within 1 year prior to screening) must agree to use a reliable method of contraception until they have completed the study and for at least 4 weeks following their final study visit. Reliable contraception is defined as a method which results in a low failure rate, i.e., less than 1% per year when used consistently and correctly, such as implants, injectables, some intrauterine contraceptive devices (IUDs), complete sexual abstinence, or a vasectomized partner. Oral contraceptive medications are allowed in this study. Female subjects who are surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) or postmenopausal (defined as no menstrual period within 1 year of screening) are also allowed to participate.

A subject who meets any of the following criteria is not eligible for participation in the study.

1. Subject with anaemia due to any cause other than iron deficiency, including, but not limited to:

   1. Untreated or untreatable severe malabsorption syndrome
   2. Immunosuppressant use. Immunosuppressants are permitted so long as there is no clinical evidence or suspicion of the immunosuppressant contributing to the subject's anaemia or affecting erythropoiesis.

   Variations to dosing are permitted at the discretion of the investigator so long as there is no clinical evidence or suspicion of the immunosuppressant contributing to the subject's anaemia or affecting erythropoiesis
2. Subject who has received prior to screening:

   1. Within 8 weeks intramuscular or intravenous (IV) iron or administration of depot iron preparation
   2. Within 2 weeks a blood transfusion
   3. Oral iron supplementation, taken specifically to treat anaemia, within the previous 4 weeks (Over the Counter (OTC) multivitamins containing iron are permitted)
3. Subjects with active inflammatory bowel disease as defined by a SCCAI score greater than 5 at Screening or a CDAI score greater than 300 in the Screening period (as assessed using the Screening haematocrit (HCT) and CDAI diary card completed by the subject for 7 days prior to planned randomization).
4. Subjects with known hypersensitivity or allergy to either the active substance or excipients of ferric maltol capsules or ferric carboxymaltose solution for IV administration
5. Subjects who have had serious adverse reactions to previous doses of ferric carboxymaltose or any other intravenous iron.
6. Subjects with contraindication for treatment with iron preparations, e.g. hemochromatosis, chronic hemolytic disease, sideroblastic anaemia, thalassemia, or lead intoxication induced anaemia.
7. Subjects with vitamin B12 or folic acid deficiency as determined by the central laboratory screening results. Subjects may start vitamin B12 or folate replacement and rescreen after at least 2 weeks.
8. Subjects who are pregnant or breast feeding.
9. Concomitant medical conditions with significant active bleeding likely to initiate or prolong anaemia.
10. Participation in any other interventional clinical study within 30 days prior to screening.
11. Subject with cardiovascular, liver, renal, haematologic, gastrointestinal, immunologic, endocrine, metabolic, or central nervous system disease that, in the opinion of the Investigator, may adversely affect the safety of the subject or severely limit the lifespan of the subject (i.e. unlikely to complete the full duration of the study).
12. Subject with significant neurologic or psychiatric symptoms resulting in disorientation, memory impairment, or inability to report accurately that might interfere with treatment compliance, study conduct or interpretation of the results (e.g., Alzheimer's disease, schizophrenia or other psychosis, active or current alcohol or drug abuse)
13. Subject who is an inmate of a psychiatric ward, prison, or other state institution.
14. Subject who is an Investigator or any other team member involved directly or indirectly in the conduct of the clinical study.
15. Subjects with severe renal impairment: creatinine clearance <30 mL/min. (Applicable to US sites Only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Mitchell, PhD, Study Director — Shield Therapeutics
Locations (44):
- United States (17):
  - Dothan, Alabama
  - Tucson, Arizona
  - Gainesville, Florida
  - Hollywood, Florida
  - Chevy Chase, Maryland
  - Saint Paul, Minnesota
  - St Louis, Missouri
  - Great Neck, New York
  - Lima, Ohio
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Beaumont, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Bountiful, Utah
  - Bellevue, Washington
  - Seattle, Washington
- Ghent, Belgium
- France (6):
  - Clichy
  - Lille
  - Lyon
  - Saint-Etienne
  - Salouël
  - Vandœuvre-lès-Nancy
- Germany (11):
  - Berlin
  - Dresden
  - Hamburg
  - Herne
  - Jena
  - Leipzig
  - Lübeck
  - Lüneburg
  - Minden
  - Oldenburg
  - Schweinfurt
- Hungary (3):
  - Budapest
  - Miskolc
  - Szeged
- Spain (6):
  - Barcelona
  - Córdoba
  - Girona
  - Madrid
  - Santiago de Compostela
  - Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 462 subjects were screened; of these, 212 subjects were not randomised (202 screening failures and 10 not assigned). 250 subjects (54% of the screened population) were randomised: 125 subjects to the ferric maltol group and 125 subjects to the IV iron group.
Groups:
- Oral Ferric Iron Compound: 30 mg capsules to be taken orally twice a day
  Ferric Maltol
- Intravenous Iron: Administered as per the local SmPC/PI
  Ferric Carboxymaltose
Period: Overall Study
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Started | 125 | 125
Received Treatment (3 pts randomised to IV were given FM instead in error. Some pts in each arm were not treated.) | 127 | 120
Completed | 93 | 106
Not Completed | 32 | 19
Not completed — Adverse Event | 10 | 2
Not completed — Lost to Follow-up | 7 | 6
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Physician Decision | 4 | 1
Not completed — Hb ≤7.5 g/dL | 0 | 2
Not completed — Blood transfusion for any reason | 0 | 1
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — TSAT above 60% or a ferritin above 800 m | 1 | 0
Not completed — None of above or not recorded | 3 | 2

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron | Total
Number analyzed (Participants) | 125 | 125 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (14.58) | 40.4 (15.54) | 40.2 (15.04)
Age, Customized [Mean (Full Range); unit: years]
  Age range | 40.0 [18 to 81] | 40.4 [19 to 77] | 40.2 [18 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 77 | 145
  Male | 57 | 48 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian/Alaskan Native | 0 | 1 | 1
  Race: Asian | 0 | 2 | 2
  Race: Black/African American | 6 | 3 | 9
  Race: White | 110 | 111 | 221
  Race: Other | 8 | 8 | 16
  Race: Native American/Pacific Islander | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 15 | 20 | 35
  Ethnicity: Not Hispanic or Latino | 99 | 94 | 193
  Ethnicity: Not Reported | 8 | 8 | 16
  Ethnicity: Unknown | 3 | 3 | 6
Fertility status (females) [Count of Participants; unit: Participants] — Population: This baseline measure is applicable to the female population only.
  Participants
    number analyzed (Participants) | 68 | 77 | 145
    Sterile | 8 | 6 | 14
    Post-menopausal | 13 | 16 | 29
    Potentially fertile | 46 | 54 | 100
    Not available | 1 | 1 | 2
Screening Hb for randomisation [Count of Participants; unit: Participants]
  <10 g/dL Female or <11 g/dL Male | 67 | 67 | 134
  ≥10 g/dL Female or ≥11 g/dL Male | 58 | 58 | 116
Baseline Hb [Count of Participants; unit: Participants]
  <9.5 g/dL | 38 | 35 | 73
  ≥9.5 g/dL | 87 | 90 | 177
IBD subgroup [Count of Participants; unit: Participants]
  Crohn's disease | 79 | 79 | 158
  Ulcerative colitis | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Either a 2g/dL Increase in Hb OR Normalization of Hb at Week 12
Description: Number of subjects achieving either a 2g/dL increase in Hb OR normalization of Hb (>=12g/dL women,>=13g/dL men) at Week 12
Time Frame: Baseline to Week 12
Population: ITT (MI)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 125 | 125
Participants
  Responder | 84 | 105
  Non-responder | 41 | 20
Statistical Analysis 1: Comparison: Oral Ferric Iron Compound vs Intravenous Iron; Test type: Non-Inferiority — A 2-sided CI for difference in the proportions of Hb responders (risk difference for ferric maltol - IV iron) between the two treatment groups, and comparing the LCL of this CI to the pre-specified non-inferiority margin of 20%. The CI was calculated using the Delta Method approach based on a logistic regression model, adjusted for treatment group, baseline Hb (below the observed median or at least the observed median), and IBD subgroup (UC or CD); p = 0.298, t-test, 2 sided; Risk Difference (RD) = -0.17, 95% CI 2-sided [-0.28 to -0.06]

2. Primary Outcome: Number of Subjects Achieving Either a 2g/dL Increase in Hb OR Normalization of Hb at Week 12
Description: Number of subjects achieving either a 2g/dL increase in Hb OR normalization of Hb (>=12g/dL women, >=13g/dL men) at Week 12
Time Frame: Baseline to Week 12
Population: re-evaluated PP
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 78 | 88
Participants
  Responder | 53 | 75
  Non-responder | 25 | 13
Statistical Analysis 1: Comparison: Oral Ferric Iron Compound vs Intravenous Iron; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.341, t-test, 2 sided; Risk Difference (RD) = -0.17, 95% CI 2-sided [-0.30 to -0.05]

3. Secondary Outcome: Change in Hb Concentration From Baseline to Week 12
Description: Change in hemoglobin concentration from baseline to Week 12.
Time Frame: Baseline to Week 12
Population: ITT (MI)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 125 | 125
g/dL | 2.45 (1.449) | 3.04 (1.576)

4. Secondary Outcome: Change in Hb Concentration From Baseline to Week 12 in Subjects With a Baseline Hb <9.5 g/dL
Description: Change in hemoglobin concentration from baseline to Week 12 in subjects with a baseline hemoglobin <9.5 g/dL.
Time Frame: Baseline to Week 12
Population: ITT (MI)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 38 | 35
g/dL | 2.83 (1.493) | 4.18 (1.686)

5. Secondary Outcome: Number of Subjects Who Experience a Change From Baseline in Hb Concentration ≥1.0 g/dL at Week 12
Description: Number of subjects who experience a change from baseline in hemoglobin concentration ≥1.0 g/dL at Week 12.
Time Frame: Baseline to Week 12
Population: ITT (MI)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 125 | 125
Participants
  Responder | 107 | 111
  Non-responder | 18 | 14

6. Secondary Outcome: Number of Subjects With Baseline Hb <9.5g/dL That Achieve an Increase in Hb Concentration of ≥1 g/dL at Week 12
Description: Number of subjects with baseline hemoglobin <9.5g/dL that achieve an increase in hemoglobin concentration of ≥1 g/dL at Week 12.
Time Frame: Baseline to Week 12
Population: ITT (MI) Not all subjects were tested.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 38 | 35
Participants
  Responder | 35 | 32
  Non-responder | 3 | 3

7. Secondary Outcome: Number of Subjects With Hb Concentration Within Normal Limits at Week 12
Description: Number of subjects with Hb concentration within normal limits at Week 12 (normal limit definition: >=12g/dL women, >=13g/dL men)
Time Frame: Baseline to Week 12
Population: ITT (MI)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 125 | 125
Participants
  Responder | 69 | 101
  Non-responder | 56 | 24

8. Secondary Outcome: Number of Subjects With Baseline Hb Concentration <9.5 g/dL That is Within Normal Limits at Week 12
Description: Number of subjects with baseline Hb concentration <9.5 g/dL that is within normal limits at Week 12 (normal limit definition: >=12g/dL women, >=13g/dL men)
Time Frame: Baseline to Week 12
Population: ITT (MI)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 38 | 35
Participants
  Responder | 12 | 28
  Non-responder | 26 | 7

9. Secondary Outcome: Proportion of Subjects Who Are Non-anaemic at 6 Months and 12 Months
Description: Long term efficacy endpoints i.e. proportion of subjects who are non-anaemic at 6 months and 12 months (normal limit definition: >=12g/dL women, >=13g/dL men)
Time Frame: Baseline to Month 6
Population: ITT (OC) Not all subjects were tested.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 125 | 125
Participants
  week 24: number analyzed (Participants) | 80 | 85
  week 24: Non-anaemic | 52 | 58
  week 24: Anaemic | 28 | 27
  week 52: number analyzed (Participants) | 61 | 56
  week 52: Non-anaemic | 37 | 36
  week 52: Anaemic | 24 | 20

10. Secondary Outcome: Change in Hb Concentration From Baseline to Week 4
Description: Change in hemoglobin concentration from baseline to Week 4.
Time Frame: Baseline to Week 4
Population: ITT (MI)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 125 | 125
g/dL | 1.27 (0.974) | 2.19 (1.133)

11. Secondary Outcome: Change in Hb Concentration From Baseline to Week 4 in Subjects With a Baseline Hb <9.5 g/dL
Description: Change in hemoglobin concentration from baseline to Week 4 in subjects with a baseline hemoglobin <9.5 g/dL.
Time Frame: Baseline to Week 4
Population: ITT (MI)
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 38 | 35
g/dl | 1.35 (0.993) | 2.99 (1.092)

12. Secondary Outcome: Number of Subjects Who Experience a Change From Baseline in Hb Concentration ≥2.0 g/dL at Week 12
Description: Number of subjects who experience a change from baseline in hemoglobin concentration ≥2.0 g/dL at Week 12.
Time Frame: Baseline to Week 12
Population: ITT (MI)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 125 | 125
Participants
  Responder | 76 | 96
  Non-responder | 49 | 29

13. Secondary Outcome: Number of Subjects With Baseline Hb <9.5g/dL That Achieve an Increase in Hb Concentration of ≥2 g/dL at Week 12
Description: Number of subjects with baseline hemoglobin <9.5g/dL that achieve an increase in hemoglobin concentration of ≥2 g/dL at Week 12.
Time Frame: Baseline to Week 12
Population: ITT (MI)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 38 | 35
Participants
  Responder | 26 | 30
  Non-responder | 12 | 5

14. Secondary Outcome: Number of Subjects Who Experience a Change From Baseline in Hb Concentration ≥1.0 g/dL at Week 4
Description: Number of subjects who experience a change from baseline in hemoglobin concentration ≥1.0 g/dL at Week 4.
Time Frame: Baseline to Week 4
Population: ITT (MI)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 125 | 125
Participants
  Responder | 75 | 105
  Non-responder | 50 | 20

15. Secondary Outcome: Number of Subjects With Baseline Hb <9.5g/dL That Achieve an Increase in Hb Concentration of ≥1 g/dL at Week 4
Description: Number of subjects with baseline hemoglobin <9.5g/dL that achieve an increase in hemoglobin concentration of ≥1 g/dL at Week 4.
Time Frame: Baseline to Week 4
Population: ITT (MI)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 36 | 33
Participants
  Responder | 22 | 31
  Non-responder | 14 | 2

16. Secondary Outcome: Number of Subjects With Hb Concentration Within Normal Limits at Week 4
Description: Number of subjects with Hb concentration within normal limits at Week 4 (normal limit definition: >=12g/dL women, >=13g/dL men)
Time Frame: Baseline to Week 4
Population: ITT (MI)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 125 | 125
Participants
  Responder | 31 | 60
  Non-responder | 94 | 65

17. Secondary Outcome: Number of Subjects With Baseline Hb Concentration <9.5 g/dL That is Within Normal Limits at Week 4
Description: Number of subjects with baseline Hb concentration <9.5 g/dL that is within normal limits at Week 4 (normal limit definition: >=12g/dL women, >=13g/dL men)
Time Frame: Baseline to Week 4
Population: ITT (MI)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 38 | 35
Participants
  Responder | 2 | 15
  Non-responder | 36 | 20

18. Secondary Outcome: Number of Subjects Who Experience a Change From Baseline in Hb Concentration ≥2.0 g/dL at Week 4
Description: Number of subjects who experience a change from baseline in hemoglobin concentration ≥2.0 g/dL at Week 4.
Time Frame: Baseline to Week 4
Population: ITT (MI)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 125 | 125
Participants
  Responder | 26 | 75
  Non-responder | 99 | 50

19. Secondary Outcome: Number of Subjects With Baseline Hb <9.5g/dL That Achieve an Increase in Hb Concentration of ≥2 g/dL at Week 4
Description: Number of subjects with baseline hemoglobin <9.5g/dL that achieve an increase in hemoglobin concentration of ≥2 g/dL at Week 4
Time Frame: Baseline to Week 4
Population: ITT (MI)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 38 | 35
Participants
  Responder | 5 | 28
  Non-responder | 33 | 7

20. Other Pre Specified Outcome: Change From Baseline Physical Component and Mental Component Score
Description: A multipurpose, proprietary health survey with 36 questions. It was constructed to survey health status in the Medical Outcomes Study and designed for use in clinical practice and research & general population surveys.
  The SF-36 includes one multi-item scale that assesses 8 health components:
  Physical Functioning Component; Social Functioning Component; Role-Physical Component; Bodily Pain Component; Mental Health Component; Role-Emotional Component; Vitality Component; & General Health Component.
  These 8 health component scales can be further summarised into 2 summary scores, the Mental Component Score & the Physical Component Score where higher values mean a better outcome.
  Both scales range from 0 to 100, where higher scores indicate better health status.
  The survey will be administered at study visits as indicated in the schedule of assessments, commencing pre-randomization at Visit 2. The survey will be completed by the subjects in their native language.
Time Frame: Baseline to Week 52 (LOCF)
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 125 | 125
score on a scale
  Physical component score | 3.0 (7.62) | 2.5 (7.52)
  Mental component score | 3.3 (8.32) | 2.6 (7.60)

21. Other Pre Specified Outcome: Number of Patients With Treatment-emergent Adverse Events (AEs)
Description: Number of Patients with Treatment-emergent Adverse Events (AEs).
Time Frame: Baseline to Week 52
Population: 3 subjects were randomised to IV iron but were given ferric maltol in error.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 127 | 120
Participants | 75 | 43

22. Other Pre Specified Outcome: Number of Patients With Treatment-emergent Serious Adverse Events (SAEs)
Description: Number of Patients with Treatment-emergent Serious Adverse Events (SAEs).
Time Frame: Baseline to Week 52
Population: 3 subjects were randomised to IV iron but were given ferric maltol in error.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
Number analyzed (Participants) | 127 | 120
Participants | 9 | 3

ADVERSE EVENTS:
Time Frame: The analysis of AEs focuses on TEAEs, which were defined as any AE that occurred on or worsened after the first dose of IMP and up to 14 days after the last dose of IMP (week 52 if study completed)
Description: The figures provided won't equal the total number of participants as several patients may have had the same AE.
  250 patients were randomised: 125 pts in the ferric maltol group & in the IV iron group each. Of these, 247 pts received at least 1 dose of IMP & were included in the safety analysis. 2 pts randomised to IV were not treated: 1 pt was randomised in error & was withdrawn, 1 pt withdrew consent; 1 pt randomised to FM was not treated & lost to follow-up; 3 pts were given FM instead of IV.
Arm/Group | Oral Ferric Iron Compound | Intravenous Iron
All-Cause Mortality (participants affected / at risk) | 1/127 | 0/120
Serious Adverse Events (participants affected / at risk) | 12/127 | 4/120
Other Adverse Events (participants affected / at risk) | 75/127 | 43/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Ferric Iron Compound (N=127) | Intravenous Iron (N=120)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3) | 2 (4)
Infections and infestations (Infections and infestations) | 3 (5) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Cardiac disorders (Cardiac disorders) | 2 (2) | 0 (0)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions (General disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Ferric Iron Compound (N=127) | Intravenous Iron (N=120)
Abdominal pain (General disorders) | 12 (13) | 15 (29)
Nausea (Gastrointestinal disorders) | 6 (8) | 2 (5)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 4 (4) | 4 (4)
Crohns disease (Gastrointestinal disorders) | 3 (3) | 4 (5)
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 4 (4) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 10 (11) | 4 (6)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 4 (4)
Asthenia (General disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 40 (69) | 15 (29) — TEAEs in <2% of Subjects Overall by SOC
Infections and infestations (Infections and infestations) | 29 (45) | 22 (32) — TEAEs in <2% of Subjects Overall by SOC
General disorders and administration site conditions (General disorders) | 9 (9) | 6 (8) — TEAEs in <2% of Subjects Overall by SOC
Nervous system disorders (Nervous system disorders) | 9 (13) | 4 (4) — TEAEs in <2% of Subjects Overall by SOC
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 9 (11) | 4 (4) — TEAEs in <2% of Subjects Overall by SOC
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 11 (11) | 2 (2) — TEAEs in <2% of Subjects Overall by SOC
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 7 (9) | 2 (2) — TEAEs in <2% of Subjects Overall by SOC
Investigations (Investigations) | 5 (6) | 2 (4) — TEAEs in <2% of Subjects Overall by SOC
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 (5) | 3 (3) — TEAEs in <2% of Subjects Overall by SOC
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (1) — TEAEs in <2% of Subjects Overall by SOC
Psychiatric disorders (Psychiatric disorders) | 4 (4) | 1 (1) — TEAEs in <2% of Subjects Overall by SOC
Eye disorders (Eye disorders) | 2 (2) | 2 (2) — TEAEs in <2% of Subjects Overall by SOC

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT02680756/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT02680756/SAP_002.pdf